CLINICAL TRIAL: NCT03164733
Title: Age Dependency of Biological Reaction on Wear Particles
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Georg Matziolis, head of the orthopaedic department, Jena University Hospital
Other Study IDs: AgeWear
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Total Hip Arthroplasty; Wear
MeSH Terms: interventions — Infectious Disease Incubation Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples of patients that have received a total hip arthroplasty
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- <40: patients younger than 40 years
  Interventions: Other: incubation
- 40-60: patients younger than 60 years and not older than 40 years
  Interventions: Other: incubation
- 60-80: patients younger than 80 years and not older than 80 years
  Interventions: Other: incubation
- >80: patients older than 80 years
  Interventions: Other: incubation

INTERVENTIONS:
Other: incubation — standardized wear particles are co-incubated with isolated patient cells (monocytes)

SUMMARY:
Wear is the main reason for revision operations after joint arthroplasty. While the survival of modern implants is often longer than the expected life span in old patients, young patients (<60 years) have to expect at least one wear induced revision operation. The reason is the throughout all registries consistantly significantly reduced implant survival rates in young patients. In the swedish arthrplasty registry the 15 year survival for patients older than 75 years is 95 % and for those younger than 50 years is 75 %. This corresponds to a 5fold increased revision rate (5 % vs. 25 %) 15 years after implantation. This significant difference cannot be explained by the higher activity of younger patients alone. Patient specific factors, that modulate the biological reaction on wear particles, are therefore highly probable. These could explain the significant age dependency of implant survival.

The main hypothesis of this study is therefore, that the biological reaction on wear particles depends on the patients age.

ELIGIBILITY:
Inclusion Criteria:

* having received a total hip arthroplasty 4 weeks before blood sample for this study

Exclusion Criteria:

* no informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients having received a total hip arthroplasty 4 weeks before blood sample for this study
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
biological reaction | one hour
  TNF-alpha concentration one hour after incubation of patient cells with wear particles in-vitro

IPD SHARING:
Plan to Share IPD: No